CLINICAL TRIAL: NCT01932060
Title: Effects of Different Oxytocin Infusions on Blood Loss and Postpartum Hemoglobin Values in Patients Undergoing Elective Cesarean Delivery
Brief Title: Oxytocin Infusions and Blood Loss in Patients Undergoing Elective Cesarean Delivery.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Alex James Butwick, Principal Investigator, Stanford University
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 28015
Record Dates: First submitted 2013-08-21; First posted 2013-08-30 (Estimated); Results first posted 2017-02-01 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-12

CONDITIONS: Postpartum Hemorrhage
Keywords: Oxytocin; blood loss; Cesarean delivery
MeSH Terms: conditions — Postpartum Hemorrhage; Hemorrhage | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxytocin Infusion 1 (Experimental): Oxytocin Infusion 15 U/hr to begin after the delivery of the fetus and to terminate at the time of patient discharge from the post-anesthesia care unit.
  Interventions: Drug: Oxytocin Infusion
- Oxytocin Infusion 2 (Active Comparator): Oxytocin infusion 2.5 U/hr to begin after the delivery of the fetus and to terminate at the time of discharge from the post-anesthesia care unit.
  Interventions: Drug: Oxytocin Infusion

INTERVENTIONS:
Drug: Oxytocin Infusion — Patient will receive a blinded infusion of oxytocin after the time of delivery of the fetus which will terminate at the time of discharge from the post-anesthesia care unit.
  Other Names: Oxytocin; Pitocin

SUMMARY:
Although prior dose-finding studies have investigated the optimal bolus dose of oxytocin to initiate adequate uterine tone, it is unclear what oxytocin infusion regimen is required to maintain adequate uterine tone after delivery. The study investigators aim to compare two different infusion rates of oxytocin to assess the optimal infusion regimen for reducing blood loss in women undergoing elective Cesarean delivery.

DETAILED DESCRIPTION:
Oxytocin (pitocin) is a drug commonly used in obstetric practice, and the drug effect is to increase the muscular tone of the uterus to reduce uterine bleeding after neonatal delivery. Pregnant patients undergoing elective (scheduled)Cesarean delivery routinely receive oxytocin after delivery of the baby. Post-delivery, oxytocin is commonly administered as an IV bolus and/or infusion. No previous studies have accurately assessed differences in oxytocin infusions after delivery in patients undergoing elective cesarean delivery. Thus the study aim is to investigate which infusion rate can optimally provide adequate maintenance of uterine tone during Cesarean delivery while being associated with minimal or no maternal side-effects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant patients with uncomplicated pregnancies:
* ASA (American Association of Anesthesiologists) class 1 or 2 patients.
* Singleton pregnancies.

Exclusion Criteria:

* ASA class 3 or 4 patients.
* Known drug allergy to intravenous oxytocin.
* Significant medical or obstetric disease.
* Known uterine abnormality.
* Known placental abnormality.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2013-08; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander J Butwick, F.R.C.A., Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children's Hospital, Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oxytocin Infusion 1 | Oxytocin Infusion 2
Started | 27 | 24
Completed | 27 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxytocin Infusion 1 | Oxytocin Infusion 2 | Total
Number analyzed (Participants) | 27 | 24 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (6) | 32 (5) | 33 (6)
Gender [Count of Participants; unit: Participants]
  Female | 27 | 24 | 51
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 24 | 51

OUTCOME MEASURES:

1. Primary Outcome: Total Estimated Blood Loss
Description: Blood loss will be measured volumetrically (based on measured volume of blood within the suction chamber) and gravimetrically (based on blood weight on blood soaked laps).
Time Frame: immediately at end of surgery
Measure: Median (Inter-Quartile Range); unit: ml
Arm/Group | Oxytocin Infusion 1 | Oxytocin Infusion 2
Number analyzed (Participants) | 27 | 24
ml | 512 [405 to 740] | 634 [340 to 886]

2. Secondary Outcome: Hemoglobin Indices After Cesarean Delivery
Description: Study investigators will assess maternal hemoglobin levels at 24hr after cesarean delivery
Time Frame: 24 hr after cesarean delivery
Measure: Median (Inter-Quartile Range); unit: g/dl
Arm/Group | Oxytocin Infusion 1 | Oxytocin Infusion 2
Number analyzed (Participants) | 27 | 24
g/dl | 11. [9.9 to 11.8] | 11.2 [10.3 to 12.2]

ADVERSE EVENTS:
Time Frame: during period of hospitalization - max 7 days
Arm/Group | Oxytocin Infusion 1 | Oxytocin Infusion 2
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/24
Other Adverse Events (participants affected / at risk) | 0/27 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No